CLINICAL TRIAL: NCT00082823
Title: An Open-Label, Long-Term, Safety and Tolerability Study of VEGF Trap Administered Intravenously in Patients With Advanced Solid Tumors or Lymphoma
Brief Title: Intravenous VEGF Trap in Treating Patients With Relapsed or Refractory Advanced Solid Tumors or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REGENERON-VGFT-ST-0304; MSKCC-03138; CDR0000360846 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Cancer
Keywords: recurrent grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; stage IV grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; recurrent adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; unspecified adult solid tumor, protocol specific; recurrent adult soft tissue sarcoma; advanced adult primary liver cancer; recurrent adult primary liver cancer; recurrent cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer; fallopian tube cancer; ovarian sarcoma; recurrent ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent endometrial carcinoma; stage IV endometrial carcinoma; recurrent uterine sarcoma; stage IV uterine sarcoma; recurrent ovarian germ cell tumor; stage IV ovarian germ cell tumor; ovarian stromal cancer; recurrent vaginal cancer; stage IVA vaginal cancer; stage IVB vaginal cancer; recurrent prostate cancer; stage IV prostate cancer; recurrent penile cancer; stage IV penile cancer; recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; recurrent bladder cancer; stage IV bladder cancer; recurrent vulvar cancer; stage IVB vulvar cancer; distal urethral cancer; proximal urethral cancer; recurrent urethral cancer; urethral cancer associated with invasive bladder cancer; primary peritoneal cavity cancer; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Neoplasms; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Sarcoma; Carcinoma, Hepatocellular; Uterine Cervical Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial; Endometrial Neoplasms; Vaginal Neoplasms; Prostatic Neoplasms; Penile Neoplasms; Testicular Neoplasms; Urinary Bladder Neoplasms; Vulvar Neoplasms; Urethral Neoplasms; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — aflibercept

INTERVENTIONS:
Biological: ziv-aflibercept

SUMMARY:
RATIONALE: Intravenous VEGF Trap may stop the growth of solid tumors or non-Hodgkin's lymphoma by stopping blood flow to the cancer.

PURPOSE: This phase I trial is studying the side effects of VEGF Trap in treating patients with relapsed or refractory advanced solid tumors or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of intravenous VEGF Trap in patients with relapsed or refractory advanced solid tumors or non-Hodgkin's lymphoma.

Secondary

* Determine the steady-state pharmacokinetics of this drug in these patients.
* Determine the ability of this drug to bind circulating vascular endothelial growth factor in these patients.
* Determine whether antibodies to this drug develop in these patients.
* Determine, preliminarily, the ability of repeated doses of this drug to alter tumor growth and vascular permeability in these patients.

OUTLINE: This is an open-label, multicenter, extension study.

Patients receive VEGF Trap* IV over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients receive the same drug dose that they received in MSKCC-03137 (VGFT-ST-0202)

Patients are followed monthly for 3 months.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 3-6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-Hodgkin's lymphoma OR primary or metastatic solid tumor located in at least one of the following sites:

  * Liver
  * Soft tissue
  * Pelvis
  * Other site that is suitable for delayed contrast-enhancing MRI
* Relapsed or refractory disease

  * Failed all conventional therapeutic options AND not amenable to existing therapeutic options
* Must have completed the active phase (through study visit 9) of MSKCC-03137 (VGFT-ST-0202) without experiencing dose-limiting toxicity
* No prior or concurrent CNS metastases (brain or leptomeningeal)

  * No new neurological symptoms during treatment on MSKCC-03137 (VGFT-ST-0202)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* No severe or uncontrolled hematologic condition

Hepatic

* Not specified

Renal

* No severe or uncontrolled renal condition

Cardiovascular

* No severe or uncontrolled cardiovascular condition

Pulmonary

* No severe or uncontrolled pulmonary condition

Other

* No severe or uncontrolled gastrointestinal, immunologic, or musculoskeletal condition
* No other medical or psychiatric condition or adverse social circumstance that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception during and for 3 months after study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent epoetin alfa, filgrastim (G-CSF), or sargramostim (GM-CSF)

Chemotherapy

* Not specified

Endocrine therapy

* No concurrent adrenal corticosteroids, except low-dose replacement therapy
* No concurrent systemic hormonal contraceptive agents

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent non-steroidal anti-inflammatory drugs, including cyclo-oxygenase-2 (COX-2) inhibitors
* No concurrent anticoagulant or antiplatelet drugs, including warfarin, heparin, or aspirin

  * Concurrent low-dose (i.e., 1 mg) warfarin for maintaining patency of venous access devices allowed
* No other concurrent standard or investigational agents for this malignancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-01; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P. Tew, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Lockhart AC, Rothenberg ML, Dupont J, Cooper W, Chevalier P, Sternas L, Buzenet G, Koehler E, Sosman JA, Schwartz LH, Gultekin DH, Koutcher JA, Donnelly EF, Andal R, Dancy I, Spriggs DR, Tew WP. Phase I study of intravenous vascular endothelial growth factor trap, aflibercept, in patients with advanced solid tumors. J Clin Oncol. 2010 Jan 10;28(2):207-14. doi: 10.1200/JCO.2009.22.9237. Epub 2009 Nov 30. PMID 19949018
- [Result] Wang-Gillam A, Tew WP, Rothenberg ML, Dupont J, Cooper W, Sternas L, Buzenet G, Sosman JA, Spriggs DR, Lockhart AC. A phase I study of subcutaneously administered aflibercept (VEGF trap) in a new formulation in patients with advanced solid tumors. Invest New Drugs. 2012 Oct;30(5):1958-61. doi: 10.1007/s10637-011-9753-y. Epub 2011 Oct 15. PMID 22002018